CLINICAL TRIAL: NCT02285530
Title: GDF15 (Growth Differentiation Factor 15) Based TPF Induction Chemotherapy for Oral Squamous Cell Carcinoma Patients at T3/T4cN0M0 Stage: a Phase II Randomized Controlled Trial
Brief Title: GDF15 Based TPF Induction Chemotherapy for OSCC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, associate professor,PHD,DDS,MD, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOSCAN
Record Dates: First submitted 2014-10-22; First posted 2014-11-07 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Mouth Neoplasms; Carcinoma, Squamous Cell
Keywords: head and neck squamous cell carcinoma, GDF15, TPF
MeSH Terms: conditions — Mouth Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPF group (Experimental): The patients in the experimental group received the TPF induction chemotherapy for 2 cycles followed by radical surgery and post-operative radiotherapy.
  docetaxel:75mg/m2 cisplatin:75 mg/m2 5-Fu:750 mg/m2/day
  Interventions: Drug: TPF induction chemotherapy; Procedure: surgery group; Radiation: Post-operative radiotherapy
- surgery group (Other): Radical resection of the primary lesion and full neck,radiotherapy was arranged 4 to 6 weeks after surgery
  Interventions: Procedure: surgery group; Radiation: Post-operative radiotherapy

INTERVENTIONS:
Drug: TPF induction chemotherapy — TPF induction chemotherapy: 2 cycles; docetaxel(75mg/m^2), cisplatin(75 mg/m^2), 5-Fu(750 mg/m^2/day) for 5 days; 16 days later, the 2nd cycle.
  Other Names: TPF protocol group
  Arms: TPF group
Procedure: surgery group — Radical resection of the primary lesion and full neck dissection(functional or radical) with proper reconstruction(pedicle or free flap) were performed.
Radiation: Post-operative radiotherapy — Radiotherapy was arranged 4 to 6 weeks after surgery. Routine external beam radiotherapy, such as conformal or intensity modulated radiotherapy was performed and the dose was 1.8-2 Gy/day, 5 days/week for 6 weeks, and totally 54-60 Gy.

SUMMARY:
The purpose of this study is to confirm the predictive value of GDF15 expression for TPF induction in T3/T4cN0M0 patients with OSCC

DETAILED DESCRIPTION:
Induction chemotherapy is regarded as an effective way to reduce or downgrade the locally advanced or aggressive cancers, and to improve the chance of eradication of the locoregional lesions by radical surgery and/or radiotherapy. However, there are still debates on the clinical value of induction chemotherapy for patients with advanced and resectable oral squamous cell carcinoma. A prospective, open label, parallel, interventional, randomized control trial on TPF induction chemotherapy indicate there is no difference in overall survival, disease free survival, local regional recurrence free survival and metastasis free survival between experimental group and control group, however, the subgroup analysis proves that the induction chemotherapy of TPF protocol could benefit the patients with GDF15 high expression and cN0 locally advanced oral squamous cell carcinoma. (Yang et al, GDF15 is a potential predictive biomarker for TPF induction chemotherapy and promotes tumorigenesis and progression in oral squamous cell carcinoma, Ann Oncol, 2014) This prospective, interventional, randomized control trial was to prove that this predictive biomarker for T3/T4cN0M0 patients with high GDF15 expression benefitting from TPF induction chemotherapy.

The patients would receive TPF induction chemotherapy followed by radical surgery and post-operative radiotherapy (the experimental group) or radical surgery and post-operative radiotherapy (the control group). The study had a power of 80% on the basis of an assumed 5-year survival rate of 85% in the experiment group and 66% in the control group, with use of a two-sided log-rank test at a level of significance of 0.05. The recruitment period would be 2 years, and the follow-up period would be 5 years, and 15% of patients would drop out early or be lost to follow-up. A maximum of 36 patients per group were to be recruited with stplan 4.5 software calculation. （Department of Biostatics, MD Anderson Cancer Center, University of Texas，USA）The patients in the experimental group received the TPF induction chemotherapy for 2 cycles followed by radical surgery and post-operative radiotherapy. The palpable edges of the primary lesion (both the longest and shortest axis) were marked before induction chemotherapy by at least four points, which were 0.5cm away. The patients in the control group received the radical surgery and post-operative radiotherapy.

Induction chemotherapy: For the patients who were randomly assigned to receive TPF induction chemotherapy, peripherally inserted central catheter was firstly inserted before intravenous infusion, docetaxel(at a dose of 75mg/m2 of body surface area) was administered as a 2-hour intravenous infusion, followed by intravenous cisplatin(75 mg/m2), administered during a period of 2 to 3 hours. Then, 5-Fu (750 mg/m2/day) was administered as a 120-hour continuous intravenous infusion for 5 days. Induction chemotherapy was given every 3 weeks for 2 cycles, unless there was disease progression, unacceptable toxic effects, or withdrawal of consent by the patients. Dexamethasone was given before docetaxel infusion to prevent docetaxel-related hypersensitivity reactions, skin toxic effects, and fluid retention; prophylactic antibiotics were also given starting on day 5 of each cycle for 3 days. Hydration with diuretic and antiemetic treatment was also performed. Primary prophylaxis with recombinant granulocyte colony-stimulating factor was not suggested. Chemotherapy dose reductions were allowed for grade 3/4 toxicities occurring after cycle 1: 25% and 50% dose reductions of the three chemotherapy agents were suggested for grade 3 and grade 4 hematologic toxicities or gastrointestinal toxicities, respectively; 25% and 50% cisplatin dose reductions were suggested for grade 3 and grade 4 renal toxicities, respectively. Surgery was performed at least 2 weeks after completion of induction chemotherapy.

Surgery: Radical resection of the primary lesion and full neck dissection(functional or radical) with proper reconstruction(pedicle or free flap) were performed. The safety margins of the primary lesion were 1.0-1.5cm far away from the palpable margins of the lesion; for patients who received induction chemotherapy, the safety margins were 1.0cm away from the marks that were placed before induction chemotherapy, to ensure the same extent surgery in both arms. Frozen sections during surgery were performed to confirm adequate margins.

Post-operative radiotherapy: Radiotherapy was arranged 4 to 6 weeks after surgery. Routine external beam radiotherapy, such as conformal or intensity modulated radiotherapy was performed, and the dose was 1.8-2 Gy(Gray)/day, 5 days/week for 6 weeks, and totally 54-60 Gy, in the patient with high risk features, such as positive surgical margin, extra capsular nodal spread, vascular embolism, concurrent chemotherapy with cisplatin 80mg/m2 was suggested.

A complete medical history was obtained and tumor assessment was performed at baseline. Clinical tumor response was assessed by clinical evaluation and imaging study and was characterized according to the criteria of response evaluation criteria in solid tumors (version 1.1) before surgery. Post-operative pathologic response was assessed by post-operative pathologic examination as good and bad response. A good response was defined as absence of any tumor cells (pathologic complete response) or presence of scattered foci of a few tumor cells (minimal residual disease with <10% viable tumor cells); otherwise, a bad pathologic response was defined. Toxic effects were assessed weekly during and after completion of induction chemotherapy and radiotherapy according to the common terminology criteria for adverse events (version 3.0).

Overall survival was calculated from the date of randomization to the date of death; disease free survival was calculated from the date of randomization to tumor recurrence or distant metastasis or death from any cause; locoregional recurrence/distant metastasis free survival was calculated from the date of randomization to locoregional recurrence/distant metastasis of tumor or death from any cause. Time to locoregional recurrence/distant metastasis was calculated from the date of finishing treatment to tumor locoregional recurrence/distant metastasis. Patients were monitored by every three months in the first two years, every six months in the next 2 years, and once a year thereafter until death or data censoring.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years old.
* Sex: both males and females.
* Karnofsky performance status (KPS) >60.
* Histological biopsy confirming squamous cell carcinoma of the oral cavity (tongue, gingiva, buccal mucosa, floor of mouth, palate, and retromolar region).
* GDF1 high expression
* Clinical stage III/IVA (T1-2, N2, M0 or T3-4, N2, M0, UICC[international Union Against Cancer ] 2002) with resectable lesions.
* Adequate hematologic function: white blood cell >3,000/mm3, hemoglobin>8g/L, platelet count>80,000/mm3.
* Hepatic function: ALAT(alanine aminotransferase)/ASAT(aspartate transaminase) <2.5 times the upper limit of normal (ULN), bilirubin <1.5 times ULN.
* Renal function: serum creatinine <1.5 times ULN.
* Written informed consent

Exclusion Criteria:

* Evidence of distant metastatic disease and other cancers.
* Surgical procedure of the primary tumors or lymph nodes (except diagnostic biopsy).
* Previous radiotherapy or chemotherapy.
* Other previous malignancies within 5 years.
* Can not tolerate the treatment protocol with systematic diseases such as history of severe pulmonary or cardiac diseases.
* Legal incapacity or limited legal capacity.
* Creatinine clearance <30ml/min.
* Pregnancy (confirmed by serum or urine β-HCG) or lactation period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 year
  2-year overall survival rate as a measure by the numbers of living patients

SECONDARY OUTCOMES:
disease free survival | 2 year
  2-year disease free survival as a measure by the number of patients without recurrence or death
local recurrence free survival | 2 year
  2-year local recurrence free survival as a measure by the number of patients without recurrence
distant metastasis free survival | 2 year
  2-year distant metastasis free survival as a measure by the number of patients without metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Ninth People's Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China